CLINICAL TRIAL: NCT01823328
Title: Ketamine Versus Etomidate for Sedation of Emergency Department Patients During Rapid Sequence Intubation
Brief Title: Ketamine Versus Etomidate for Rapid Sequence Intubation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR 13-3601
Record Dates: First submitted 2013-03-28; First posted 2013-04-04 (Estimated); Results first posted 2019-05-24 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Airway Control; Anesthesia; Intubation; Complication
Keywords: Intubation; Airway; Emergent intubation; Rapid sequence intubation; Rapid sequence induction; RSI; Ketamine; Etomidate; Sepsis; Sedative; Sedation
MeSH Terms: conditions — Sepsis | interventions — Ketamine; Etomidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): Subjects in the ketamine arm will receive ketamine for sedation prior to rapid sequence intubation (RSI).
  Interventions: Drug: Ketamine
- Etomidate (Active Comparator): Subjects in the etomidate arm will receive etomidate for sedation prior to rapid sequence intubation (RSI).
  Interventions: Drug: Etomidate

INTERVENTIONS:
Drug: Ketamine — Subjects will receive ketamine for sedation prior to rapid sequence intubation.
  Other Names: Ketanest; Ketaset; Ketalar
  Arms: Ketamine
Drug: Etomidate — Subjects will receive etomidate for sedation prior to rapid sequence intubation.
  Other Names: Amidate
  Arms: Etomidate

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of ketamine and etomidate during rapid sequence intubation (RSI).

DETAILED DESCRIPTION:
This study is a randomized controlled trial of etomidate versus ketamine during rapid sequence intubation (RSI). RSI refers to the process by which patients who require emergency airway management undergo sedation and paralysis prior to insertion of an endotracheal tube(airway tube). Patients who require intubation will be randomized to have intubation performed with either ketamine or etomidate. All other care will be at the discretion of the treating physicians. The purpose of this study is to compare the efficacy and safety of ketamine and etomidate during rapid sequence intubation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Undergoing rapid sequence intubation (RSI) in the Emergency Department

Exclusion Criteria:

* Known contraindication to ketamine or etomidate
* Patient has a condition in which an increase in heart rate or blood pressure would be hazardous, as judged by the treating physician
* Patient is known or suspected of having increased intracranial pressure, based on the history and physical examination performed by the treating physician.
* Females of child-bearing age, defined as 18-50 years, who do not have a documented pregnancy test in this institution confirming that they are not pregnant or who do not have a confirmed surgical procedure preventing pregnancy, i.e., tubal ligation, hysterectomy. The timing of the pregnancy test at which the investigative team will consider a subject to be non-pregnant is a documented negative test during current hospitalization or upon direct transfer from outside institution during current illness.
* Patient declines participation in the trial by wearing a bracelet marked "KvE declined"
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Driver, MD, Principal Investigator — Hennepin County Medical Canter
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 14 patients withdrew consent.
Period: Overall Study
Arm/Group | Ketamine | Etomidate
Started | 70 | 73
Completed (The number of completions is lower than the number started because of withdrawal by patients.) | 62 | 67
Not Completed | 8 | 6
Not completed — Withdrawal by Subject | 8 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Etomidate | Total
Number analyzed (Participants) | 62 | 67 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (20) | 49 (19) | 49 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 23 | 48
  Male | 37 | 44 | 81
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 3 | 9
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 18 | 36
  White | 38 | 37 | 75
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: SOFA Score
Description: *Maximum SOFA score within three hospital days: all patients. SOFA score is the Sequential Organ Failure Assessment. The minimum score is 0, the maximum score is 24, with higher scores indicating higher likelihood of worse outcome.
Time Frame: up to 3 days
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 62 | 67
units on a scale | 6.5 [5 to 9] | 7 [5 to 9]

2. Secondary Outcome: Mortality in Sepsis and Septic Shock
Description: Evaluate mortality for the sub-group diagnosed with sepsis and septic shock, defined as:
  - Suspected infection, and at least 2 of 4 systemic inflammatory response syndrome (SIRS) criteria:
  1. Temperature >38C or <36C
  2. Respiratory Rate >20 or PaCO2 <32 mmHg
  3. Heart Rate >90
  4. White blood cell count >12,000 or <4,000, or > 10% bands
  Septic shock:
  defined as sepsis plus either: 1) Systolic blood pressure <90 after 1L of intravenous fluid or 2) lactate >=4mmol/L
Time Frame: 30 Days
Population: Subgroup of those with sepsis
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 9 | 16
Participants | 1 | 4

3. Secondary Outcome: Number of Patients With First-pass Success
Description: The rate of first pass success, defined as successful tracheal intubation on the first attempt. An attempt is defined as the insertion and subsequent removal of the laryngoscopic device from the patient's mouth, regardless of whether an endotracheal tube was inserted.
Time Frame: up to 5 minutes (average time frame)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 62 | 67
Participants | 59 | 60

4. Secondary Outcome: Doses of Post-intubation Sedation
Description: The number of bolus doses of sedative administered post-intubation will be compared up to 6 hours (including morphine, dexmedetomidine, propofol , etomidate, ketamine, lorazepam (Ativan), midazolam (Versed), diazepam (Valium), fentanyl, hydromorphone (Dilaudid)). Infusions of these medications will be recorded separately but will not be part of this outcome.
Time Frame: up to 6 hours
Measure: Median (Inter-Quartile Range); unit: bolus doses of sedation
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 62 | 67
bolus doses of sedation | 1 [0 to 2] | 1 [0 to 2]

5. Secondary Outcome: Number of Patients With Post-intubation Hypoxemia
Description: The following will be compared between the two groups:
  * Hypoxemia and severe hypoxemia in the peri-intubation period. Peri-intubation hypoxemia was defined as during after the 5 minutes immediately after intubation.
  * Hypoxemia within the first 2 hours intubation
  Hypoxemia is defined as SpO2 less than 90%. Severe hypoxemia is defined as SpO2 less than 90% for 60 seconds or more.
Time Frame: up to 2 hours
Population: Those with oxygen saturation data
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 59 | 66
Participants
  Peri-intubation hypoxemia | 8 | 13
  Hypoxemia within 2 h of ICU admission | 1 | 5

6. Secondary Outcome: Number of Patients With Hypotension
Description: The following will be compared between the two groups:
  * Hypotension in the ED post-intubation
  * Hypotension within the first 6 hours of the hospital stay, including time spent in the ED
  Hypotension is defined as a systolic blood pressure less than 90 mm Hg
Time Frame: up to 6 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 62 | 67
Participants
  Hypotension in the first 6 hours of hospitalizatio | 24 | 30
  Hypotension in the ED | 16 | 17

7. Secondary Outcome: Peak and Plateau Pressure
Description: The Peak and plateau pressures will be compared between the two groups, with a pre-defined subgroup analysis of patients who are being intubated for severe asthma and chronic obstructive pulmonary disease (COPD). The ventilator was used to measure these values.
Time Frame: up to 30 minutes (average time frame)
Population: Those with peak and plateau pressure available
Measure: Median (Inter-Quartile Range); unit: cm water
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 60 | 65
cm water
  Peak pressure | 25 [23 to 30] | 26 [22 to 31]
  Plateau Pressure | 16 [14 to 20] | 17 [16 to 20]

8. Secondary Outcome: Mortality
Description: Mortality will be assessed at 30 days or at discharge from the hospital, whichever occurs first. This study is not powered to detect a significant difference in mortality, however; this will primarily be a safety study comparing the use ketamine versus etomidate as sedative agents for rapid sequence intubation (RSI) in the Emergency Department (ED).
Time Frame: 30 Days or Discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine | Etomidate
Number analyzed (Participants) | 62 | 67
Participants | 8 | 15

ADVERSE EVENTS:
Arm/Group | Ketamine | Etomidate
Serious Adverse Events (participants affected / at risk) | 1/62 | 0/67
Other Adverse Events (participants affected / at risk) | 0/62 | 0/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=62) | Etomidate (N=67)
Severe hypertension (Cardiac disorders) | 1 (1) | 0 (0) — After ketamine administration one patient had severely elevated blood pressure > 200/100 mm Hg

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No